CLINICAL TRIAL: NCT06078839
Title: Nafamostat Mesilate in the Treatment of Severe Infection-associated Coagulopathy: a Multicenter Randomized Controlled Trial
Brief Title: Nafamostat Mesilate in the Treatment of Severe Infection-associated Coagulopathy
Acronym: NMSICRCT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xu Li (Other)
Collaborators: Tianjin Third Central Hospital (Other); Tianjin Medical University General Hospital (Other); Shanxi Provincial People's Hospital (Other Government); Shanxi Bethune Hospital (Other); Hohhot First Hospital (Unknown); Jilin University (Other); Northern Jiangsu People's Hospital (Other); The Affiliated Hospital of Nantong University (Unknown); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital of Suzhou Medical (Unknown); Anhui Provincial Hospita (Unknown); Zhejiang Hospital (Other); Zhejiang Provincial People's Hospital (Other); The First Affiliated Hospital of Ningbo (Unknown); The First Affiliated Hospital of Wenzhou (Unknown); The Jiangxi Provincial People's Hospital (Unknown); First Affiliated Hospital of Gannan Medical University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); LanZhou University (Other); The First Affiliated Hospital of Xinjiang (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); Tongji Medical College of Huazhong University (Unknown); The Second Hospital University of South China (Other); The Fourth Affiliated Hospital of China Medical (Unknown); The First Affiliated Hospital of Liaoning (Unknown); Genertec Liaoyou Gem Flower Hospital (Unknown); The Tenth People's Hospital of Shenyang (Unknown); The Sixth People's Hospital of Shenyang (Other); Dalian NO.3 People's Hospital (Unknown); Benxi Cental Hospital (Other); Liaoyang City Central Hospital (Unknown); Huludao central hospital (Unknown)
Responsible Party: Sponsor-Investigator, Xu Li, Professor, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AF-0G-03-1.1-02
Record Dates: First submitted 2023-09-20; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Sepsis; Sepsis-induced Coagulopathy; Nafamostat Mesilate
MeSH Terms: conditions — Sepsis | interventions — nafamostat; Glucose

STUDY DESIGN:
Intervention Model Description: Nafamostat mesilate treatment group (experimental group) : Basic treatment + Nafamostat mesilate 2.0 mg/kg/d Placebo control group: Basic treatment + 5% glucose with Nafamostat mesilate equal volume
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo control group (Placebo Comparator)
  Interventions: Drug: 5% glucose
- Nafamostat mesilate treatment group (experimental group) (Experimental)
  Interventions: Drug: Nafamostat mesilate

INTERVENTIONS:
Drug: Nafamostat mesilate — Nafamostat mesilate treatment group was dissolved with 5% glucose at the dosage of 2.0mg/kg/ day to a total of 50ml(Maximum concentration 10mg/ml)
  Arms: Nafamostat mesilate treatment group (experimental group)
Drug: 5% glucose — Add 50ml of 5% glucose into a 50ml syringe
  Arms: Placebo control group

SUMMARY:
The objective of this study was to evaluate the therapeutic effect of nafamostat mesilate on patients with severe infection-related coagulation。

ELIGIBILITY:
Inclusion Criteria:

* meets the criteria for sepsis 3.0".
* Targeted population for SIC anticoagulant therapy（http://research-kudo-prediction.s3-website-ap-northeast-1.amazonaws.com/）

Exclusion Criteria:

* Age less than 18, pregnant women, and lactating women
* Patients with a history of hypersensitivity to nafamostat mesilate (previous use of nafamostat mesilate resulted in significant bleeding complications)
* Fibrinogen < 1.5g/L
* Patients with bleeding or high bleeding risk Patients in the acute phase of trauma or with active bleeding (such as flail chest, significant contusions of the lungs, liver, kidneys, spleen, retroperitoneal bleeding, pelvic fractures, etc.) History of severe traumatic brain injury, intracranial surgery, stroke, cerebral aneurysm, or arteriovenous malformation within the past month prior to enrollment Patients with a history of congenital bleeding disorders (such as hemophilia) Patients with underlying fulminant hepatitis, decompensated cirrhosis, or other severe liver diseases
* Patients receiving the following medications Patients who have received heparin and heparin analogs (including low molecular weight heparin, dalteparin, etc.) within the past 12 hours prior to treatment Patients who have received warfarin within the past 7 days prior to the study and have an INR level above normal Patients who have undergone thrombolytic therapy within the past 3 days prior to the study Patients who have received platelet inhibitors (such as aspirin, clopidogrel, ticlopidine, dipyridamole, etc.) within the past 7 days prior to the study Patients currently receiving other novel anticoagulant medications (such as Xa factor inhibitors like apixaban, rivaroxaban, edoxaban, etc., direct thrombin inhibitors like dabigatran
* ICU treatment time is expected to be no more than 24h
* Patients who have undergone cardiopulmonary resuscitation within the past 7 days prior to the study
* Patients who have participated in other studies within the 30 days prior to enrollment
* Due to irreversible disease states, such as advanced malignant tumors or other end-stage diseases; or patients in a terminal state deemed by the physician to be approaching death

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality in ICU | 7 days

SECONDARY OUTCOMES:
Improvement in organ function (SOFA score) | 7 days
DIC score (JAAM/ISTH score) changes; | 7 days
28-day all-cause fatality rate | 28-day
Adverse event rate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Xu Li, Phd, Principal Investigator — First Hospital of China Medical University

REFERENCES:
- [Derived] Yang H, Feng J, Ma Y, Ma X, Li X; EASNMS investigators. Efficacy and safety of nafamostat mesilate for sepsis (EASNMS): study protocol for a multicenter randomized controlled trial. Trials. 2025 Jul 29;26(1):262. doi: 10.1186/s13063-025-08979-4. PMID 40731293